CLINICAL TRIAL: NCT02765802
Title: A Phase 2 Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of Pegylated Interferon Lambda Monotherapy in Patients With Chronic Hepatitis Delta Virus Infection (LIMT)
Brief Title: A Study to Evaluate Pegylated Interferon Lambda Monotherapy in Patients With Chronic Hepatitis Delta Virus Infection
Acronym: LIMT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eiger BioPharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EIG-LMD-001
Record Dates: First submitted 2016-05-05; First posted 2016-05-09 (Estimated); Results first posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-12

CONDITIONS: Hepatitis D, Chronic
MeSH Terms: conditions — Hepatitis D, Chronic | interventions — peginterferon lambda-1a

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lambda 180 μg (Experimental): Lambda 180 μg once weekly, administered by subcutaneous (SC) injection, for a total of 48 weeks.
  Interventions: Drug: Peginterferon Lambda-1A
- Lambda 120 μg (Experimental): Lambda 120 μg once weekly, administered by subcutaneous (SC) injection, for a total of 48 weeks.
  Interventions: Drug: Peginterferon Lambda-1A

INTERVENTIONS:
Drug: Peginterferon Lambda-1A
  Other Names: Lambda

SUMMARY:
To evaluate safety and tolerability of lambda over a 48-week treatment period in HDV patients.

DETAILED DESCRIPTION:
Lambda is the pegylated form of interferon lambda-1a (IFN-λ), a conjugate of recombinant human interleukin 29 (rIL-29) and a linear polyethylene glycol (PEG) chain. IFN-λ and interferon alpha (IFN-α) share the common interferon (IFN)-stimulated gene induction pathway that leads to broad-spectrum antiviral activities. Since IFN-α has demonstrated anti-hepatitis delta virus (HDV) activity in patients with chronic hepatitis delta (CHD), it is postulated that pegylated IFN-λ could also induce HDV ribonucleic acid (RNA) decline in patients with CHD. Based on IFN-λ's more limited receptor distribution and previous data from studies involving treatment with IFN-λ in patients with hepatitis B virus (HBV) or hepatitis C virus (HCV), it is postulated that Lambda treatment could be associated with fewer adverse effects than IFN-α treatment. This Phase II study is designed as randomized, open-label study of Lambda 120 or 180 μg subcutaneous (SC) injection weekly for 48 weeks in patients with chronic HDV infection, and the primary objectives of the study are as follows:

* To evaluate the safety and tolerability of treatment with 2 dose levels of Lambda over a 48-week treatment period.
* To evaluate the effect of treatment with 2 different doses of Lambda on HDV RNA levels.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HDV infection of at least 6 months' duration documented by a positive HDV antibody (Ab) test, detectable and quantifiable HDV RNA by qPCR at study entry
* Serum alanine aminotransferase (ALT) > upper limit of the normal range (ULN) and <10 × ULN at screening
* Electrocardiogram (ECG) demonstrating no acute ischemia or clinically significant abnormality and a QT interval corrected for heart rate (QTcF) <450 ms for male patients and <460 ms for female patients
* Thyroid-stimulating hormone (TSH) and/or free T4 within 0.8 to 1.2 × ULN, or adequately controlled thyroid function as assessed by the investigator.
* Dilated retinal examination ≤1 year before screening
* Female patients of childbearing potential and male patients with partners of childbearing potential must agree to use adequate methods of contraception during the study and through 90 days after the last dose of study medication

Exclusion Criteria:

General Exclusions:

* Participation in a clinical trial with or use of any investigational agent within 30 days before screening, or treatment with interferons (IFNs) or immunomodulators within 12 months before screening
* Previous use of Lambda. Patients who previously participated in a clinical trial of Lambda but are confirmed to have received placebo or other non-Lambda IFNs are allowed.
* History or evidence of any intolerance or hypersensitivity to IFNs or other substances contained in the study medication.
* Female patients who are pregnant or breastfeeding. Male patients must confirm that their female sexual partners are not pregnant.

Exclusions Based on Disease

* Current or previous history of decompensated liver disease (Child-Pugh Class B or C)
* Co-infected with human immunodeficiency virus (HIV) or hepatitis C virus (HCV)
* Past history or current evidence of decompensated liver disease, defined as any of the following at screening:

  1. Bilirubin level ≥ 2.5 mg/dL unless due to Gilbert's disease
  2. Serum albumin level <3.5 g/dL
  3. International normalized ratio (INR) ≥1.5
  4. Alpha fetoprotein ≥100 ng/mL
* Evidence of significant portal hypertension; current presence or history of variceal bleeding, ascites requiring diuretics or paracentesis, or hepatic encephalopathy
* Any of the following abnormal laboratory test results at screening:

  1. Platelet count <90,000 cells/mm^3
  2. White blood cell count <3,000 cells/mm^3
  3. Absolute neutrophil count <1,500 cells/mm^3
  4. Hemoglobin <11 g/dL for women and <12 g/dL for men
  5. Serum creatinine concentration ≥1.5× ULN
  6. Confirmed creatinine clearance (CrCl) < 50 mL/min by Cockcroft-Gault
* Evidence of another form of viral hepatitis or another form of liver disease
* History of hepatocellular carcinoma
* Patients with any of the following:

  1. Current eating disorder or alcohol abuse
  2. Excessive alcohol intake
  3. In the opinion of the investigator, an alcohol use pattern that will interfere with study conduct
  4. Drug abuse within the previous 6 months before screening, with the exception of cannabinoids and their derivatives
* Prior history or current evidence of any of the following:

  1. Immunologically mediated disease
  2. Retinal disorder or clinically relevant ophthalmic disorder
  3. Any malignancy within 5 years before screening
  4. Cardiomyopathy or significant ischemic cardiac or cerebrovascular disease.
  5. Chronic pulmonary disease
  6. Pancreatitis
  7. Severe or uncontrolled psychiatric disorder
  8. Active seizure disorder
  9. Bone marrow or solid organ transplantation
* Other significant medical condition that may require intervention during the study

Exclusions Based on Concurrent Medication Use

* Therapy with an immunomodulatory agent
* Use of telbivudine
* Current use of heparin or Coumadin
* Received blood products within 30 days before study randomization
* Use of hematologic growth factors within 30 days before study randomization
* Systemic antibiotics, antifungals, or antivirals for treatment of active infection other than HBV within 14 days before study randomization
* Any prescription or herbal product that is not approved by the investigator
* Long-term treatment (> 2 weeks) with agents that have a high risk for nephrotoxicity or hepatotoxicity unless it is approved by the medical monitor
* Receipt of systemic immunosuppressive therapy within 3 months before screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Apelian, MD, PhD, MBA, Study Director — Eiger BioPharmaceuticals
Locations (4):
- Israel (2):
  - Soroka Medical Center, Beersheba
  - Shaare Zedek Medical Center, Jerusalem
- Auckland City Hospital, Grafton, Auckland, New Zealand
- The Aga Khan University and Hospital, Karachi, Pakistan

REFERENCES:
- [Background] Kotenko SV, Gallagher G, Baurin VV, Lewis-Antes A, Shen M, Shah NK, Langer JA, Sheikh F, Dickensheets H, Donnelly RP. IFN-lambdas mediate antiviral protection through a distinct class II cytokine receptor complex. Nat Immunol. 2003 Jan;4(1):69-77. doi: 10.1038/ni875. Epub 2002 Dec 16. PMID 12483210
- [Background] Sheppard P, Kindsvogel W, Xu W, Henderson K, Schlutsmeyer S, Whitmore TE, Kuestner R, Garrigues U, Birks C, Roraback J, Ostrander C, Dong D, Shin J, Presnell S, Fox B, Haldeman B, Cooper E, Taft D, Gilbert T, Grant FJ, Tackett M, Krivan W, McKnight G, Clegg C, Foster D, Klucher KM. IL-28, IL-29 and their class II cytokine receptor IL-28R. Nat Immunol. 2003 Jan;4(1):63-8. doi: 10.1038/ni873. Epub 2002 Dec 2. PMID 12469119
- [Background] Wedemeyer H, Manns MP. Epidemiology, pathogenesis and management of hepatitis D: update and challenges ahead. Nat Rev Gastroenterol Hepatol. 2010 Jan;7(1):31-40. doi: 10.1038/nrgastro.2009.205. PMID 20051970

RESULTS

PARTICIPANT FLOW:
Groups:
- Lambda 180 μg: Lambda 180 μg once weekly, administered by subcutaneous (SC) injection, for a total of 48 weeks.
  Peginterferon Lambda-1A
- Lambda 120 μg: Lambda 120 μg once weekly, administered by subcutaneous (SC) injection, for a total of 48 weeks.
  Peginterferon Lambda-1A
Period: Overall Study
Arm/Group | Lambda 180 μg | Lambda 120 μg
Started | 14 | 19
Completed | 14 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Peginterferon Lambda-1A 180 μg: Peginterferon Lambda-1A (Lambda) 180 μg once weekly, administered by subcutaneous (SC) injection, for a total of 48 weeks.
- Peginterferon Lambda-1A 120 μg: Peginterferon Lambda-1A (Lambda) 120 μg once weekly, administered by subcutaneous (SC) injection, for a total of 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Peginterferon Lambda-1A 180 μg | Peginterferon Lambda-1A 120 μg | Total
Number analyzed (Participants) | 14 | 19 | 33
Age, Continuous [Mean (Full Range); unit: years] | 43.8 [23 to 63] | 36.6 [20 to 63] | 39.7 [20 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 7 | 15 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 19 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 11 | 15
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 0 | 1 | 1
  White | 8 | 5 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Israel | 8 | 6 | 14
  Pakistan | 4 | 11 | 15
  New Zealand | 2 | 2 | 4
log HDV RNA [Mean (Full Range); unit: log IU/mL] | 3.86 [0.5 to 7.3] | 4.15 [0.5 to 6.1] | 4.03 [0.5 to 7.3]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HDV Viral Load.
Description: To evaluate the safety and tolerability of treatment with 2 dose levels of Lambda over a 48 week treatment period.
  To evaluate the effect of treatment with 2 different doses of Lambda on hepatitis D virus (HDV) ribonucleic acid (RNA) levels.
Time Frame: Week 48 (end of treatment)
Measure: Mean (Standard Deviation); unit: Change in HDV RNA log IU/mL
Arm/Group | Lambda 180 μg | Lambda 120 μg
Number analyzed (Participants) | 14 | 19
Change in HDV RNA log IU/mL | -2.14 (1.81) | -1.16 (2.38)

2. Secondary Outcome: Change From Baseline in HDV Viral Load
Description: To evaluate the proportion of patients with undetectable HDV RNA 24 weeks after the end of treatment
Time Frame: Week 72 (end of follow-up)
Measure: Mean (Standard Deviation); unit: Change in HDV RNA log IU/mL
Arm/Group | Lambda 180 μg | Lambda 120 μg
Number analyzed (Participants) | 14 | 19
Change in HDV RNA log IU/mL | -1.70 (1.70) | -0.66 (1.57)

3. Secondary Outcome: Number of Patients With a Durable Virologic Response
Description: Durable Virologic Response (DVR) = below the limit of quantitation in HDV RNA at 24 weeks post-treatment
Time Frame: Week 72
Measure: Count of Participants; unit: Participants
Groups:
- Peginterferon Lambda-1A 180 μg: Patients chronically infected with HDV who are randomized to the Peginterferon Lambda-1A 180 μg arm
- Peginterferon Lambda-1A 120 μg: Patients chronically infected with HDV who are randomized to the Peginterferon Lambda-1A 120 μg arm
Arm/Group | Peginterferon Lambda-1A 180 μg | Peginterferon Lambda-1A 120 μg
Number analyzed (Participants) | 14 | 19
Participants | 5 | 3

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected on or after the first Lambda injection, through 24 weeks post-treatment, an average of 72 weeks.
Description: Based on specific management guidelines for occurrence of Grade 3 AEs and events including hepatobiliary laboratory abnormalities, patients were allowed to interrupt treatment, dose reduce, and/or discontinue Lambda treatment during study. The dose reduction plan allowed patients who were randomized to the Lambda 180 mcg dose to receive Lambda 120 mcg or 80 mcg during study, and patients who were randomized to the Lambda 120 mcg dose to receive Lambda 80 mcg during study.
Arm/Group | Lambda 180 μg | Lambda 120 μg
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/19
Serious Adverse Events (participants affected / at risk) | 2/14 | 5/19
Other Adverse Events (participants affected / at risk) | 14/14 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lambda 180 μg (N=14) | Lambda 120 μg (N=19)
jaundice (Hepatobiliary disorders) | 2 (3) | 4 (6)
Drug-Induced Liver Injury (DILI) (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lambda 180 μg (N=14) | Lambda 120 μg (N=19)
Jaundice (Hepatobiliary disorders) | 2 | 4
Alanine Aminotransferase (ALT) increase (Investigations) | 5 | 3
Aspartate Aminotransferase (AST) Increase (Investigations) | 5 | 2
Blood bilirubin increased (Investigations) | 4 | 2
gamma-glutamyl transferase (GGT) increased (Investigations) | 2 | 2
international normalized ratio (INR) increased (Investigations) | 1 | 2
Neutrophil count decreased (Investigations) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4
Dizziness (Nervous system disorders) | 3 | 1
Dysgeusia (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 12 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritis (Skin and subcutaneous tissue disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2
Diarrhea (Gastrointestinal disorders) | 5 | 5
Dyspepsia (Gastrointestinal disorders) | 7 | 6
Nausea (Gastrointestinal disorders) | 5 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 2 | 1
Chills (General disorders) | 3 | 5
Fatigue (General disorders) | 8 | 3
Feeling cold (General disorders) | 1 | 2
Influenza like illness (General disorders) | 1 | 4
Injection site erythema (General disorders) | 5 | 1
Injection site pain (General disorders) | 5 | 1
Injection site pruritis (General disorders) | 5 | 2
Pyrexia (General disorders) | 7 | 8
Urinary tract infection (Infections and infestations) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT02765802/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT02765802/SAP_001.pdf